CLINICAL TRIAL: NCT01058018
Title: Phase II Multi-center, Double-blind, Randomized, Parallel Group, Placebo-controlled Clinical Trial for Dose-finding and Safety Study of RVX000222 in Subjects With Stable Coronary Artery Disease
Brief Title: Clinical Trial for Dose Finding and Safety of RVX000222 in Subjects With Stable Coronary Artery Disease
Acronym: ASSERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVX222-CS-005
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: Cholesterol; High density lipoprotein; Atherosclerosis; ApolipoproteinA1; Stable angina artery disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — apabetalone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A - 100 mg per day RVX000222 (Experimental): Arm A: Treatment with RVX000222 at 50 mg twice daily for 12 weeks, orally with meals in the morning and in the evening, 10 to 12 hours apart.
  Interventions: Drug: RVX000222
- B - 200 mg per day RVX000222 (Experimental): Arm B: Treatment with RVX000222 100 mg twice daily for 12 weeks, orally with meals in the morning and in the evening, 10 to 12 hours apart.
  Interventions: Drug: RVX000222
- C - 300 mg per day RVX000222 (Experimental): Arm C: Treatment with RVX000222 150 mg twice daily for 12 weeks, orally with meals in the morning and in the evening, 10 to 12 hours apart.
  Interventions: Drug: RVX000222
- D - Placebo (Placebo Comparator): Arm D: Treatment with placebo for 12 weeks, orally with meals in the morning and in the evening, 10 to 12 hours apart.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RVX000222 — RVX000222 twice a day for 12 weeks
  Other Names: RVX-208; apabetalone
  Arms: A - 100 mg per day RVX000222; B - 200 mg per day RVX000222; C - 300 mg per day RVX000222
Drug: Placebo — Placebo twice a day for 12 weeks
  Arms: D - Placebo

SUMMARY:
The purpose of this study is to investigate dose range, safety and efficacy of RVX000222 in subjects with stable coronary artery disease.

DETAILED DESCRIPTION:
One-third of the US population, almost 80 million adults, have cardiovascular disease and mortality associated with heart disease still remains as a leading cause of death around the world. The major risk factors for cardiovascular disease associated with atherosclerosis is dyslipidemia, characterized by high levels of low density lipoprotein (LDL) and/or low levels of high density lipoprotein (HDL). The widespread use of statins in patients at risk for cardiovascular disease has led to lower LDL levels but has had little effect on HDL levels. HDL has a well established role in atherosclerosis and cardiovascular disease protection. HDL mediates the removal of cholesterol from the atherosclerotic plaques for elimination from the body. The cardioprotective component of HDL consists of apolipoprotein A1 (ApoA1). Recent intervention studies with synthetic HDL particles and recombinant ApoA1 have shown that HDL has the capacity to reverse coronary atherosclerosis. Increasing ApoA1 is likely to have a favorable effect on atherosclerotic plaque size and stability, and on cardiovascular diseases. RVX000222 is a member of a novel class of small molecules that are candidates for the treatment of dyslipidemia by increasing plasma levels of HDL through increased ApoA1 transcription.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years of age.
2. If female, non-pregnant (as determined by a negative serum pregnancy test at Screening), non-lactating, and not of childbearing-potential or willing to practice acceptable form of birth control. If male, be willing to practice an acceptable form of birth control.
3. Documented coronary artery disease such as stable angina, coronary artery bypass graft, myocardial infarction within the past 90 days, or a history of percutaneous coronary intervention greater than 90 days before randomization
4. Taking a stable dose of statin therapy for at least 30 days prior to enrollment into the study with, in the investigators opinion, an unlikely need for statin dose adjustment during the course of the study.
5. Have given signed informed consent to participate in this study

Exclusion Criteria:

1. A female who is pregnant or lactating?
2. Participated in any research study, or been on an investigational drug within the last 30 days?
3. Currently have any of the following Illnesses:

   * Heart disease needing surgical repair
   * Coronary Artery bypass surgery in the last 90 days
   * PCI or Stent placement in the last 90 days
   * Left Ventricular ejection fraction
   * Evidence of cardiac electrophysiologic instability
   * Renal Impairment
   * Uncontrolled Hypertension 160/95 (2 consecutive Measurements)
   * Triglycerides ≥ 400 mg/dl (at Screening)
   * Liver: Total bilirubin > ULN, ALT/AST 1.5 > ULN at Screening
   * History of Drug or Alcohol abuse in last 12 months
   * History of Malignancy ≤ 5 years
4. Currently taking any immunosuppressant's
5. Any changes in stain therapy doses in last 30 days
6. Use of Fibrates at any dose
7. Use of Niacin ≥ 250 mg per day
8. Have any medical or surgical condition which might significantly alter the absorption, distribution, metabolism or excretion of medication including but not limited to any of the following: cholecystitis, Crohn's disease or ulcerative colitis?
9. Have any surgical or medical condition which in the opinion of the Investigator may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study?
10. Using other investigational drugs and devices at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer?
11. Have a history of noncompliance to medical regimens or unwillingness to comply with the study protocol?
12. Have any condition that in the opinion of the investigator would confound the evaluation and interpretation of efficacy and/or safety data?
13. Directly involved in the execution of this study?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The percent change in ApoA1 from baseline to 12 weeks post-randomization for each treatment arm compared to placebo. | from baseline to 12 weeks post-study drug treatment

SECONDARY OUTCOMES:
Compare the dose and time response relationships for major lipids (ApoA1, total cholesterol, HDL-C, LDL-C, non-HDL-C, TG, ApoB, LDL, and HDL-subclasses) over 4, 8 and 12 weeks time course. | 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steve Nicholls, MD, PhD, Principal Investigator — Intravascular Ultrasound Core Lab, Clevelend Clinic
Locations (1):
- Orange County Research Center, Tustin, California, United States

REFERENCES:
- [Derived] Nicholls SJ, Gordon A, Johansson J, Wolski K, Ballantyne CM, Kastelein JJ, Taylor A, Borgman M, Nissen SE. Efficacy and safety of a novel oral inducer of apolipoprotein a-I synthesis in statin-treated patients with stable coronary artery disease a randomized controlled trial. J Am Coll Cardiol. 2011 Mar 1;57(9):1111-9. doi: 10.1016/j.jacc.2010.11.015. Epub 2011 Jan 20. PMID 21255957